CLINICAL TRIAL: NCT05585489
Title: Individualization of Music-based Cueing During Gait in Parkinson's Disease. An Exploratory Cross-over Trial
Brief Title: Individualization of Music-based Cueing During Gait in Parkinson's Disease.
Acronym: MUSIGAIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Emilie Hutin, Research engineer, Henri Mondor University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A00959-32
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Gait Disorders, Neurologic; Parkinson Disease
MeSH Terms: conditions — Gait Disorders, Neurologic; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with moderate idiopathic Parkinson's disease (Experimental)
  Interventions: Other: Gait training with musical cue

INTERVENTIONS:
Other: Gait training with musical cue — Entraînement de 20 minutes de marche à vitesse confortable sur un parcours ovale de 20 mètres au laboratoire ARM avec la technique d'indiçage musical personnalisé de la longueur de pas.

SUMMARY:
Spatio-temporal correction of the step is a key component of gait rehabilitation in Parkinson's disease. Walking rehabilitation techniques using visual or auditory cueing of the cadence or step length have been tested to prevent or correct the lack of consistency of the step. An auditory cue of the duration of the step, encouraging it to be extended according to patient own capacities during gait has been proposed. The cue is integrated into music and is presented in an open-loop approach.

The present study aimed to evaluate the effect of the individual music-based cueing of the step length on gait in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Idiopathic Parkinson's disease based on UKPDSBB criteria
* 10-meter walking comfortable speed between 0,30 and 1,10 m/s
* Capacities to walk with shoes during at least 20 minutes without assistance
* Signature of informed consent

Exclusion Criteria:

* Non-affiliation to Social Security
* Person under protection (e.g. under protection of justice)
* Auditory disorders without treatment
* Cognitive disorders that limit the understanding of the study according to the medical investigator
* Other neurological or orthoêdic disorders that addect walking
* Participating in another Category 1 or 2 interventional clinical study for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Step length | Before and just after the intervention (day 1)
  Step length during confortable gait over 8 meters

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire Analyse et Restauration du Mouvement, Créteil, France

IPD SHARING:
Plan to Share IPD: No